CLINICAL TRIAL: NCT03835845
Title: An Observational, Prospective Multicentre Clinical Study to Assess the Safety and Clinical Performance of a New Single-use Negative Pressure Wound Therapy System (PICO 7Y) for the Simultaneous Management of Bilateral Closed Incisions in Oncoplastic Breast Surgery Patients
Brief Title: A Clinical Study to Assess the Safety and Clinical Performance of a New Dressing (PICO7Y) in Breast Surgery Patients
Acronym: PICO7Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1704P7Y
Record Dates: First submitted 2019-01-07; First posted 2019-02-11 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Oncoplastic Breast Surgery; Bilateral Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PICO7Y (Experimental): PICO 7Y is a single-use NPWT System consisting of a small portable pump & pump clip, 2 AA batteries, 2 large multisite dressings, 2 extension tubes and secondary fixation strips.
  Interventions: Device: PICO7Y

INTERVENTIONS:
Device: PICO7Y — The PICO 7Y pump maintains NPWT at -80 mmHg (nominal) to two wound surfaces simultaneously. Exudate is managed by the dressings through a combination of absorption and evaporation of moisture through the outer film. The PICO 7Y kit is intended to be used for up to 7 days on low exuding wounds. For moderately exuding wounds the system is intended to be used for up to 4 days without a dressing change. For 7 days use on moderately exuding wounds additional dressings will be supplied.

SUMMARY:
The purpose of the study is to assess the use of a wound dressing system called PICO7Y following a two-sided breast surgery. PICO7Y is a new dressing system made to treat two incisions/wounds at the same time, and the purpose of this study is to check how the dressing is working by looking at data on how well the dressing performs while you wear it and to check if doctors and patients are happy with it.

PICO7Y is based on another dressing called PICO.

DETAILED DESCRIPTION:
It is thought that Negative Pressure Wound Therapy may have numerous mechanisms of action when used to manage surgical incisions, including reducing oedema, stimulating perfusion and managing exudate. Post-operative oedema in the peri-wound tissue is thought to limit tissue perfusion and high levels of wound fluid loss have been correlated with increased risk of post-operative infection and dehiscence23. Application of NPWT to the closed wound has been reported to improve patient comfort through reduced dressing changes and to lessen the period during which post-operative fluid discharges from the incision. Xia et al (2014)24 demonstrated that in 20 patients with infected wounds, NPWT resulted in significantly increased blood flow in the wounds when compared to pre application levels. In a study by Young et al (2013)25 four patients with pressure ulcers had oedema and wound bed thickness assessed during follow-up. They demonstrated a rapid reduction of peri-wound tissue oedema over four days and a 20% increase in the thickness of the wound bed by seven days of therapy.

Risk factors such as smoking and obesity have shown to increase complications follow oncoplastic surgery26 and it is possible that such populations could benefit more from the application of the NPWT. Furthermore there are a number of bilateral or multi wound indications where provision of a single device with the Y connection may represent a cost saving to the healthcare system. However, ultimately the use of NPWT for oncoplastic breast surgery closed incisions will be judged on whether it can increase the healing success rate while minimising complications. Holt and Murphy (2015)27 assessed the use of PICO single use NPWT system when applied to 24 patients with closed incisions following therapeutic resection. The contralateral breast underwent simultaneous symmetrising breast reduction with standard care dressings applied allowing for direct comparison. Although the cohort was too small to draw meaningful statistical conclusions they noted a lower incidence of wound breakdown (4.2% vs. 16.7%) and shorter time to healing (10.7 days vs. 16.1 days) in the NPWT group. However, this difference was partly attributed to the more extensive and complex nature of the therapeutic surgery. Similarly in a category of patients undergoing breast surgery with primary wound closure, Pellino et al (2014)19 showed significantly lower surgical site events when treated with PICO.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have understood and provided written informed consent (reference section 9.1)
* Female subjects who must be at least eighteen (18) years of age.
* Willing and able to make all required study visits.
* Able to follow instructions.
* Subjects must be undergoing, at the same time, both an oncoplastic breast surgery and a symmetrising breast reduction on the contralateral breast and have closed incisions that would benefit from NPWT.
* Subjects whose incisions will fit comfortably within the area of the pad of the dressing sizes provided.

Exclusion Criteria:

* Contraindications (per the PICO 7Y IFU) or hypersensitivity to the use of the investigational product or their components (i.e., silicone adhesives and polyurethane films [direct contact with wound], acrylic adhesives [direct contact with skin], polyethylene fabrics and super-absorbent powders [polyacrylates]) within the dressing.
* Subjects with skin features (e.g. tattoos, skin colour, pre-existing scarring) which in the opinion of the Investigator, will interfere with the study assessments.
* Suspected or confirmed allergy to any of the components of the ancillary products should they be deemed required, e.g. in the case of SECURA No-sting barrier skin wipes for patients with fragile skin.
* Subjects with a local infection, close or at the site of the incision, at the time of surgery
* Subjects with incisions that are actively bleeding unless haemostasis has been achieved.
* Subjects with a genetic or acquired disease capable of negatively impact the closed incision healing.
* Subjects with a history of poor compliance with medical treatment.
* Subjects who have participated previously in this clinical trial.
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.
* Individuals from vulnerable populations including pregnant women and adult females over 75 years.
* Subjects who have received adjuvant chemotherapy within the last 30 days prior to surgery.
* Patients who at the end of the surgery have only one breast operated.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Clinical performance PICO 7Y NPWT system within 7 days of surgery | within 7 days of surgery
  To assess clinical performance of the PICO 7Y NPWT system through its capacity to deliver negative pressure consistently at -80 mmHg, to both the reconstructed breast and the contralateral breast, during a period of 7 days. This will be measured by assessing the incision wound on Day 7, using CDC wound assessment criteria. Photographs will also be taken of the incision wound with treatment and after treatment.
Clinical performance PICO 7Y NPWT system | within 14 days of surgery
  To assess clinical performance of the PICO 7Y NPWT system through its capacity to deliver negative pressure consistently at -80 mmHg, to both the reconstructed breast and the contralateral breast, during a period of 7 days. This will be measured by assessing the incision wound on Day 14 using CDC wound assessment criteria. Photographs will also be taken of the incision wound with treatment and after treatment.
Clinical performance PICO 7Y NPWT system within 30 days of surgery | within 30 days of surgery
  To assess clinical performance of the PICO 7Y NPWT system through its capacity to deliver negative pressure consistently at -80 mmHg, to both the reconstructed breast and the contralateral breast, during a period of 7 days. This will be measured by assessing the incision wound on Day 30, using CDC wound assessment criteria. Photographs will also be taken of the incision wound with treatment and after treatment.
Safety of the PICO7Y NPWT system through number of Adverse Events, Device Deficiencies and Serious Adverse Events. | 1 year
  Safety will be assessed by reporting any Adverse Events or Device deficiencies, and any Serious adverse events.

SECONDARY OUTCOMES:
Rate of successful healing at day 30 | up to Day 30
  via photographs of the wound incision taken at Day 0, Day 14, and Day 30
Clinician Acceptability | 1 year
  Assessed with the electronic Case Report Forms, questioning the clinician's acceptability of the device
Patient Acceptability | 1 year
  Assessed with the electronic Case Report Forms, questioning the patient's acceptability of the device
Ease of Application | 1 year
  Assessed with electronic Case Report Forms, questioning ease of application as well as questionnaires given to the participants.
Comfort | up to Day 7
  Assessing patient comfort during wear by measuring the Visual Analogue Score at day 0 and day 7.
Ease of Removal | 1 year
  Assessed with electronic Case Report forms, questioning ease of removal as well as questionnaire.
Dressing Wear Time | 1 year
  Assessed with electronic Case Report Forms as well as patient-facing questionnaires.
Incidence of Surgical Site Complications | up to Day 30
  This will be measured by assessing the incision wound with CDC criteria at Day 0 to Day 30.
Evaluate change in health-related quality of life | up to Day 30
  Assessed by using EQ-5D 5L questionnaires at Day 0, Day 14 and Day 30.

CONTACTS AND LOCATIONS:
Overall Officials: John Murphy, MBChB, Principal Investigator — Oncoplastic Breast Surgeon; Brian Gilchrist, PhD, Study Chair — Smith & Nephew - Global Clinical Strategy
Locations (5):
- Academic Hospital Maastricht, Maastricht, Netherlands
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Free Hospital, London
  - Whythenshawe Hospital, Manchester
  - Nottingham Breast Institute, Nottingham